CLINICAL TRIAL: NCT05178628
Title: The Impact of Thromboprophylaxis on Progression Free Survival of Patients With Advanced Pancreatic Cancer: The Pancreatic Cancer & Tinzaparin Prospective (imPaCT-PRO) Study
Brief Title: The Impact of Thromboprophylaxis on Progression Free Survival of Patients With Advanced Pancreatic Cancer
Acronym: imPaCT-PRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michalis Karamouzis (Other)
Responsible Party: Sponsor-Investigator, Michalis Karamouzis, Prof. Michalis Karamouzis, Institute of Molecular Medicine and Biomedical Research
Organization: Institute of Molecular Medicine and Biomedical Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: imPaCT-PRO-01
Record Dates: First submitted 2021-12-15; First posted 2022-01-05 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Pancreatic Cancer; Thromboembolism
Keywords: Thromboprophylaxis; Advanced Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Thromboembolism | interventions — Tinzaparin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, multicenter, open-label, blinded-endpoint Phase III clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with Innohep® and chemotherapy (Experimental): The patients in this arm will receive Innohep and chemotherapy with Gemcitabine + Nab-Paclitaxel (NabG) as per clinical practice.
  Interventions: Drug: Innohep
- Patients treated with chemotherapy (Active Comparator): The patients in this arm will receive chemotherapy with Gemcitabine + Nab-Paclitaxel (NabG) as per clinical practice.
  Interventions: Drug: Chemotherapy: Gemcitabine + Nab-Paclitaxel

INTERVENTIONS:
Drug: Innohep — Patients will receive Tinzaparin sodium 20.000 Anti-Xa IU/ml in prefilled syringes. Administered at 175 Anti-Xa IU/Kgr of body weight, subcutaneously, once daily
  Other Names: Tinzaparin sodium
  Arms: Patients treated with Innohep® and chemotherapy
Drug: Chemotherapy: Gemcitabine + Nab-Paclitaxel — All patients will receive chemotherapy per clinical practice
  Arms: Patients treated with chemotherapy

SUMMARY:
This is a prospective, randomized, multicenter, open-label, blinded-endpoint Phase III clinical trial to investigate the impact of thromboprophylaxis using innohep, beyond anticoagulation in the improvement of the clinical outcomes in active pancreatic cancer patients receiving systemic anti-neoplasmatic treatment. The number of patients that will be enrolled is 450. The enrollment period is 24 months and the follow up period is 10 months.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) has the worst prognosis of any malignancy. Venous thromboembolism (VTE) occurs in 1:5 PC patients and is associated with significantly reduced progression-free survival (PFS). Phase III randomised controlled trials concluded that targeted thromboprophylaxis with low molecular weight heparins (LMWH) resulted in an 82% reduction in the relative risk of VTE without increasing major bleeding events, and that 11 patients were needed to be treated to prevent one VTE during chemotherapy. The benefits observed in the many of reported studies could not be accounted for by VTE prevention alone. Numerous experimental studies have demonstrated the antitumour, anti-metastatic and chemo-resistance reversal effect of LMWH.

The vast majority of the so far published evidence assessing the efficacy and safety of VTE prevention in ambulatory cancer patients is based on mixed patient populations with various types of cancers. Thus, current studies do not allow to estimate the real effect of long-term prophylaxis on clinical outcomes in selected homogeneous high-thrombotic risk patients.

An approach more specific to PC and restricted to advanced or metastatic patients is a modern and attractive strategy to assess the benefit of thromboprophylaxis in VTE prevention and beyond anticoagulation.

The objective of the imPaCT-PRO trial is to investigate the impact of thromboprophylaxis beyond anticoagulation in the improvement of the clinical outcomes in active PC patients receiving systemic anti-neoplasmatic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced or metastatic PC (confirmed by the recommended histological and imaging methods).
2. Age ≥ 18 years.
3. Planning to start 1st line chemotherapy with NabG.
4. Eastern Cooperative Group (ECOG) 0-2.
5. Life expectancy >6 months.
6. Written informed consent.

Exclusion Criteria:

1. Subjects with contraindication to receive anticoagulant:

   1. Any hypersensitivity to anticoagulant or excipients.
   2. History of heparin-induced thrombocytopenia type II (HIT II).
   3. Active major bleeding or pre-diathesis for major bleeding
   4. Septic endocarditis.
2. Creatinine clearance <20 mL/min according to Cockcroft-Gault formula.
3. Platelet count < 50 G/L at inclusion.
4. Hepatic dysfunction defined as at least one of the following: AST and/or ALT > 5 x ULN, bilirubin > 2 x ULN.
5. Recent (< 1 month) oncological surgery, major abdominal or thoracic surgery, major orthopedic surgery, vascular surgery.
6. Recent (< 1 month) acute coronary syndrome or any other arterial thrombosis, thrombotic or hemorrhagic stroke.
7. Patients on chronic anticoagulation or on dual anti-platelet treatment.
8. Pregnancy/lactation or insufficient contraception during the study and up to 3 months after the study.
9. Severe concomitant disease that as per investigator's judgement is not compatible with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS of patients | 12 months
  PFS of patients receiving thromboprophylaxis with tinzaparin, in comparison with the PFS of patients not receiving such prevention
The number of VTE events during the trial | 12 months
  All objectively confirmed VTE events during the study per treatment arm including symptomatic distal deep vein thrombosis (DVT), symptomatic or incidental proximal DVT (including iliac and cava thrombosis), symptomatic or incidental pulmonary embolism (PE) or both DVT and PE (co-primary endpoint) or fatal PE or vein thrombosis of rare localisation (i.e., splanchnic vein or cerebral vein thrombosis).

SECONDARY OUTCOMES:
% of patients experiencing at least one major bleeding event | Through study completion, an average of 2 years
  % of patients experiencing at least one major bleeding event, according to the International Society on Thrombosis and Haemostasis (ISTH) criteria during the study per treatment arm.
% of patients experiencing any bleeding event | Through study completion, an average of 2 years
  % of patients experiencing any bleeding event, including major, clinically relevant non-major bleeding (CRNMB) and minor bleeding events during the study per treatment arm.
VTE events | Through study completion, an average of 2 years
  Incidence of VTE events, per event type, during the study per treatment arm
Patients with complete or partial response | Through study completion, an average of 2 years
  ORR, defined as the percentage of patients with complete response (CR) or partial response (PR) based on RECIST criteria
Change from baseline in QoL | at 4 and 10 months
  Change from baseline in QoL at 4 months and 10 months per treatment arm. QoL will be determined with the EORTC QLQ-C30 version 3.0. and EORTC QOL-PAN26 questionnaires according to the corresponding scoring manual

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Institute of Molecular Medicine and Biomedical Research, Athens, Attica
  - Eygenideio Hospital, Oncology Department, Athens, Attica

IPD SHARING:
Plan to Share IPD: No